CLINICAL TRIAL: NCT07319897
Title: A Prospective, Multicenter, Diagnostic Study Evaluating 68Ga-BCMA PET/CT for Targeting BCMA Expression in Multiple Myeloma.
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: The First Hospital of Jilin University (Other); The Second Hospital of Hebei Medical University (Other); Beijing Anzhen Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PFBC01
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Multiple Myeloma and Malignant Plasma Cell Neoplasms; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: multiple myeloma; bcma; PET/CT; diagnosis; multicenter
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-BCMA PET/CT (Experimental): Every patient will receive 68Ga-BCMA PET/CT
  Interventions: Diagnostic Test: 68Ga-BCMA PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-BCMA PET/CT — Intravenous administration of the investigational BCMA-targeted radiopharmaceutical, followed by a whole-body PET/CT scan performed per a standardized protocol.

SUMMARY:
This is a prospective, multicenter, diagnostic imaging study designed to evaluate the diagnostic performance and clinical utility of BCMA-targeted Positron Emission Tomography/Computed Tomography (PET/CT) in patients with multiple myeloma and other palsma cell disorders. The study aims to non-invasively visualize and quantify the whole-body biodistribution of BCMA expression.

ELIGIBILITY:
Inclusion Criteria:

(1) patients with suspected or previously diagnosed multiple myeloma (MM) who were scheduled for bone marrow aspiration or tissue biopsy within two weeks, including those undergoing initial diagnostic evaluation or follow-up/re-evaluation for disease monitoring or relapse; (2) patients with confirmed symptomatic MM; (3) ability to understand and voluntarily sign written informed consent; (4) ability to comply with study procedures; and (5) Eastern Cooperative Oncology Group (ECOG) performance status ≤2.

Exclusion Criteria:

pregnancy or lactation; inability to comprehend study procedures or cooperate with protocol requirements; or any other condition judged by the investigator to potentially interfere with study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of 68Ga-BCMA PET/CT | From enrollment to the end of PET/CT at 4 weeks
  To determine the diagnostic accuracy of BCMA PET/CT for detecting active myeloma lesions, using biopsy confirmation as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Kang, M.D, Ph.D, Principal Investigator — Peking University First Hospital; Yujun Dong, M.D, Ph.D, Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Beijing An Zhen Hospital of the Capital University of Medical Sciences, Beijingcun, Hebei
  - Beijing Tsinghua Changgung Hospital, Beijingcun, Hebei
  - Peking University First Hospital, Beijingcun, Hebei
  - the Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - First Hospital of Jilin University, Jilin, Jilin

IPD SHARING:
Plan to Share IPD: Undecided
The current approved protocol and informed consent forms do not include provisions for broad sharing of individual participant data with external researchers. The data generated are complex, integrating sensitive clinical information with novel imaging biomarkers, and require significant resources to prepare for responsible sharing. Data may be available for collaborative research upon reasonable request to the Principal Investigator, subject to execution of appropriate data transfer and use agreements.

REFERENCES:
- [Result] Song L, Jiang S, Yang Q, Huang W, Qiu Y, Chen Z, Sun X, Wang T, Wu S, Chen Y, Zeng H, Wang Z, Kang L. Development of a Novel Peptide-Based PET Tracer [68Ga]Ga-DOTA-BP1 for BCMA Detection in Multiple Myeloma. J Med Chem. 2024 Sep 12;67(17):15118-15130. doi: 10.1021/acs.jmedchem.4c00759. Epub 2024 Aug 21. PMID 39167092
- [Result] Wang T, Yang Q, Huang W, Sun X, Lei Y, Xu H, Song L, Duan X, Liu F, Wang W, Bao Z, Gao J, Wang F, Kang L. Development and Preclinical Validation of a Novel 89Zr-Labeled BCMA-Targeting Antibody for ImmunoPET Imaging: Application in Multiple Myeloma Models and First-In-Nonhuman-Primates. J Med Chem. 2025 Jul 24;68(14):14843-14858. doi: 10.1021/acs.jmedchem.5c01010. Epub 2025 Jun 25. PMID 40558019
- [Result] Gu T, Chen Z, Wang T, Dong Y, Kang L. B-cell maturation antigen targeted PET/CT imaging in multiple myeloma: a first-in-human study. J Hematol Oncol. 2025 Nov 14;18(1):101. doi: 10.1186/s13045-025-01758-3. PMID 41239440